CLINICAL TRIAL: NCT01850173
Title: Effects of Whole Body Vibration Training in Severe Chronic Obstructive Pulmonary Disease Patients
Brief Title: Whole Body Vibration in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Eulogio Pleguezuelos, Doctor, Hospital de Mataró
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAT-VIB01
Record Dates: First submitted 2013-05-02; First posted 2013-05-09 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- static work with a vertical vibration platform (Experimental): The training was designed to perform static work of the lower limbs. Patients worked in a squatting position, with 30º of hip flexion and 55º of knee flexion, holding onto the bars of the WBV platform.
  Interventions: Device: A vertical vibration platform Fitybe
- Control group (No Intervention): general recommendations about physical activity and lifestyle

INTERVENTIONS:
Device: A vertical vibration platform Fitybe — They performed 6 series, and each series consisted of four 30-second repetitions with a frequency of 35 Hz and 2 millimeters of amplitude, with 60 seconds of rest between each series.
  Arms: static work with a vertical vibration platform

SUMMARY:
The investigators designed the current study with the main objective of determining whether Whole Body Vibration Training (WBVT) alone improves muscular force and/or modifies the functional capacity parameters in severe Chronic Obstructive Pulmonary Disease (COPD) patients referred to a rehabilitation programme.

ELIGIBILITY:
Inclusion Criteria:

* severe COPD defined as a post-bronchodilator forced expiratory volume at one second (FEV1)/ forced vital capacity (FVC) < 0.7 and FEV1 < 50% predicted,
* stable disease defined as no exacerbation,
* hospital admission or change in treatment in the previous 3 months.

Exclusion Criteria:

* other significant respiratory disease (bronchiectasis,
* lung fibrosis, asthma, etc),
* active smoking,
* severe cardiovascular,
* neurological, and/or metabolic pathology that could interfere with the results,
* total hip, knee or ankle arthroplasty,
* previous vitreous haemorrhage,
* severe alcoholism (> 80 g/day) and
* severe malnutrition (BMI < 19 Kg/m2) to reduce the risk of falling and dropouts.

Ages: 55 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
isokinetic knee flexor and extensor testing muscular force | basal, 3 months follow up
  the change between basal - and 3 months follow up.
distance performed in the six minutes walking test (6MWT) | Basal, 3 months follow up
  the change between basal - and 3 months follow up.

SECONDARY OUTCOMES:
respiratory muscular strength was assessed with maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) | Basal, 3 month follow up
  the change between basal - and 3 months follow up.

OTHER OUTCOMES:
Complications | 3 months follow up
  cardiac events, increase in respiratory symptoms, knee pain during whole body vibration training.

CONTACTS AND LOCATIONS:
Overall Officials: Eulogio Pleguezuelos, PhD, Principal Investigator — Hospital de Mataró
Locations (1):
- Eulogio Pleguezuelos, Mataró, Barcelona, Spain

REFERENCES:
- See also: Hospital de Mataró. Consorci Sanitari del Maresme — http://www.csdm.cat